CLINICAL TRIAL: NCT06921070
Title: Usage and Adverse Events of Physical Restraints in an Intensive Care Unit - an Observational Cohort Study
Brief Title: Usage and Adverse Events of Physical Restraints in an Intensive Care Unit
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00057; am23Sutter
Record Dates: First submitted 2025-03-18; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Physical Restraints
Keywords: Intensive Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this retrospective observational single-center cohort study is to (1) examine the frequency of physical restraint use in a Swiss intensive care unit, (2) identify related adverse events, and (3) determine risk factors associated with their use and complications in critically ill adult patients.

DETAILED DESCRIPTION:
Physical restraints are widely used in intensive care units (ICU) worldwide to protect patients by preventing them from removing medical devices, accidentally taking out breathing tubes (self-extubation), or falling. However, while they are intended to keep patients safe, restraints can also have negative effects. Their use may increase agitation, self-extubation, infections, blood clots, longer hospital stays, and even a higher risk of death. Studies have also linked physical restraints to long-term problems, such as cognitive decline and post-traumatic stress disorder. However, most studies lack strong evidence and cannot exclude the influence of other factors.

This retrospective observational single-center cohort study aims to:

1. Determine the frequency with which physical restraints are used in a Swiss ICU
2. Identify the type and frequency of adverse events associated with physical restraint use
3. Identify other factors linked to physical restraints use and specific complications during intensive care of critically ill adult patients.

Furthermore, the study examines the use of chemical sedation with physical restraint use and the risk of delirium.

The results of this study will help improve patient care and contribute to better guidelines for physical restraint use in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e., patients ≥18 years of age)
* Being physically restrained in the intensive care unit at the University Hospital Basel between 2010 and 2023

Exclusion Criteria:

* Patients younger than 18 years.
* Patients with documented refusal to use data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all consecutive adult patients (i.e. >= 18 years of age) being physically restrained in the intensive care unit at the University Hospital Basel between 2010 and 2023.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient demographics | 2010-2023
  Demographic information (e.g. age, sex) is collected to assess potential associations with physical restraint use.
Acute prehospital management data | 2010-2023
  Data from acute prehospital management, as documented in emergency medical services (EMS) treatment protocols, is collected
Duration of ICU stay | 2010-2023
  The length of ICU stay is recorded.
Duration of hospital stay | 2010-2023
  The length of the total hospital stay is recorded.
Discharge destination | 2010-2023
  The destination at discharge is recorded.
Date of physical restraint use | 2010-2023
  The specific date of physical restraint use to each patient is documented.
Reason for physical restraint use | 2010-2023
  The documented reason for applying physical restraints, as recorded in nursing and physician progress notes, is analyzed.
Type of physical restraints used | 2010-2023
  The specific type of physical restraints used to patients during ICU stay is recorded.
Restraint Duration | 2010-2023
  To characterize the restraint period, the duration of the physical restraint period is collected from the patient record in the hospital file.
Level of consciousness at onset of restraint | 2010-2023
  To characterize the restraint period, the patient's level of consciousness at the onset of physical restraint is collected from the patient record in the hospital file.
Clinical neurologic monitoring score | 2010-2023
  A score from validated neurological assessment tool (e.g., RASS, SAS, GCS, ICDSC, STESS) is recorded during the ICU stay. The specific tool used, as well as the scale of the score and meaning behind the score, depends on the neurological assessment documented in the patient register.
Critical illness severity score | 2010-2023
  Disease severity is assessed using a standardized scoring system recorded in the patient register, such as APACHE II, SAPS II, and SOFA. The specific scoring system used depends on the clinical documentation available. The scale of the score and meaning behind the score depends on the severity assessment that has been applied.
Charlson Comorbidity Index | 2010-2023
  The Charlson Comorbidity Index (CCI) is calculated based on pre-existing comorbidities and additional diagnoses. The CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. It assigns weighted scores (from 0 to maximal 6) to 17 comorbid conditions (e.g., heart disease, diabetes, cancer), resulting in a total score ranging from 0 to 33, if the patient had the most severe form of each of the 17 conditions.
Laboratory parameters | 2010-2023
  Routine laboratory value for e.g. CRP, albumin, LDH, CK, procalcitonin, white blood cell levels, creatinine, liver enzymes, blood gas analyses, and metabolic data, is collected. The specific parameters recorded may vary depending on the laboratory assessments documented in the patient register. All values will be reported using their respective units of measurement.
Complications associated with physical restraint use | 2010-2023
  The complication occurring during or after physical restraint use, including infections, shock, hemorrhage, ischemia, hypoxia, arrhythmia, cardiopulmonary arrest, and organ failure, is recorded.
Glasgow Outcome Score | 2010-2023
  The Glasgow Outcome Score (GOS) is calculated based on the assessment of key clinical outcomes such as in-hospital mortality, survival, survival with neurofunctional alteration, return to premorbid neurological function, and hospital readmission to determine the patient outcome.
  The GOS ranges from 1 (death) to 5 (good recovery).
Therapeutic intervention | 2010-2023
  The therapeutic intervention is document based on the data available in the patient register. This includes information on treatment duration, dosage and number of treatment medication, number of neuroleptic, sedative and analgesic drugs, invasive procedures, such as intubation, mechanical, ventilation, vasopressors, installation of central lines, nutrition, etc. The specific interventions recorded depend on the clinical documentation available. All reported values will follow their respective units of measurement.
Vital signs | 2010-2023
  Vital signs are analyzed based on the data available in the patient register. These may include blood pressure, heart rate, respiratory rate, oxygen saturation, body temperature, and level of consciousness. The specific parameters recorded depend on the clinical documentation available. All values will be reported using their respective units of measurement. The collected parameters are aggregated to provide an overall assessment of the patient's clinical condition.
Fluid balance data | 2010-2023
  Fluid balance data, including the administration of fluids such as blood products, crystalloids, and enteral/parenteral nutrition, are documented
Diagnostic procedure | 2010-2023
  The diagnostic procedure (invasive or non-invasive) during intensive care, such as radiologic imaging, lumbar puncture, etc. and restraint usage during such diagnostic procedures is documented.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof. Dr. med., Principal Investigator — University Hospital Basel, Clinic for Intensive Care Medicine
Locations (1):
- University Hospital Basel, Clinic for Intensive Care Medicine, Basel, Canton of Basel-City, Switzerland